CLINICAL TRIAL: NCT02775318
Title: Efficacy Of Ultrasound Guided Stellate Ganglion Block To Relieve Vasospasm Following Clipping Of Cerebral Aneurysm
Brief Title: Stellate Ganglion Block Using Ultrasound Guidance For Treatment Of Post Clipping Cerebral Vasospasm
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, NAVNEH SAMAGH, Senior Resident In Neuroanesthesia,Department of Anesthesia and Intensive Care, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NK/1286/DM/1060
Record Dates: First submitted 2016-05-09; First posted 2016-05-17 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Cerebral Vasospasm
Keywords: Stellate Ganglion; Digital Subtraction Angiography; Transcranial Doppler Ultrasonography
MeSH Terms: conditions — Vasospasm, Intracranial | interventions — Bupivacaine; Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stellate Ganglion Block (Other): After diagnosis of vasospasm patients were administered ultrasound guided Stellate Ganglion block using 10 cc of 0.5% Inj Bupivacaine on the same side of vasospasm or the side contralateral to the focal neurological deficit.Patients were then assessed using transcranial Doppler and digital subtraction angiography after 30 minutes
  Interventions: Procedure: Stellate Ganglion Block; Drug: Bupivacaine; Procedure: Transcranial Doppler; Procedure: Digital Subtraction Angiography

INTERVENTIONS:
Procedure: Stellate Ganglion Block — Under aseptic conditions, transducer is placed on the surface of the neck at the level of C6 vertebrae. The internal jugular vein, carotid artery, thyroid gland, trachea, C6 vertebrae, transverse process of C6, esophagus , longus colli with its covering prevertebral fascia and esophagus are visualized. A 25-gauge Quincke spinal needle was inserted paratracheal towards the middle of the longus colli muscle. The endpoint of the injection was the ultrasound image of the tip of the needle as it penetrates the prevertebral fascia covering the longus colli muscle. The drug is then injected and spread of drug is visualized in real time.
Drug: Bupivacaine — 10 ml of 0.5% injection bupivacaine is used for giving stellate ganglion block on the side of cerebral vasospasm
  Other Names: Sensorcaine; Marcaine
Procedure: Transcranial Doppler — The principle on which the TCD works is that with arterial narrowing, the blood flow velocity within the vessel increases. A good correlation has been found between the TCD blood flow velocities and vasospasm. The MCA velocity greater than 120 cm/sec indicates mild vasospasm , velocity greater than 130 cm/sec indicates moderate vasospasm and velocity greater than 200 cm/sec indicates severe vasospasm.
Procedure: Digital Subtraction Angiography — Digital subtraction angiography is a direct method for the assessment of vessel caliber. It generates high resolution, high contrast and low artifact images using digital subtraction technology. Direct visualization using DSA is the gold standard for the radiographic diagnosis of cerebral vasospasm
  Other Names: DSA

SUMMARY:
The present study has been designed to assess the efficacy and safety of Stellate Ganglion Block (SGB) in relieving symptomatic cerebral vasospasm following aneurysmal clipping. The effect was assessed by both Digital Subtraction Angiography(DSA) and Transcranial Doppler (TCD).

DETAILED DESCRIPTION:
Anesthesiologist was informed about the patients (Post clipping for cerebral aneurysm) having neurological deterioration (hemiparesis, aphasia, apraxia, hemianopia, or neglect), or a decrease of ≥ 2 points on the Glasgow Coma Scale(GCS) and in whom the duration of symptoms lasted for at least 1 hour. Anesthesiologist was also informed if increased cerebral blood flow velocity was found on routine daily Transcranial Doppler(TCD) evaluation of such patients. A cerebral Computed tomography(CT) scan was performed at this time to rule out ventricular dilation or any other focal brain lesion explaining the clinical symptoms. In such patient Central venous pressure(CVP) was maintained at 8-10 mm of Hg and systolic blood pressure was maintained between 160-200 mm Hg (using infusion of vasopressors such as phenylephrine or dopamine if required). Oral/ nasogastric nimodipine (60 mg 4 hourly) was continued and hemoglobin was maintained at ≥ 10 gm/dl.

Diagnosis Of Vasospasm By Transcranial Doppler A 2 megahertz (MHz) transcranial Doppler ultrasound probe was used to insonate vessels through the temporal acoustic window. Extracranial Internal Carotid Artery (ICA) was insonated in the neck using a linear probe of 8- 13 MHz. Using Transcranial Doppler (TCD) probe, a tracing of waveform of Middle Cerebral Artery (MCA) was identified and confirmed using standard criteria. Peak Systolic Velocity and Mean Flow Velocity were assessed. Pulsatility Index and Resistivity Index were assessed. LINDEGAARD ratio was calculated.

Diagnosis Of Vasospasm By Digital Subtraction Angiography (DSA) Patients were shifted to Digital subtraction Angiography room and an emergency cerebral angiographic study was performed using Philips Allura Xper FD20/10 machine. Vasospasm was diagnosed on DSA and the vessel diameter was measured at the mid A1 segment of Anterior cerebral artery(ACA) and mid M1 segment of Middle Cerebral Artery (MCA). Vasospasm was classified as mild (<25%), moderate (25% to 50%), or severe (>50%) with respect to two - dimensional diameter at the mid A1 and mid M1 segment of ACA and MCA respectively. Location of vasospasm was classified as unilateral vs bilateral, single vessel involvement vs multiple vessel involvement or diffuse vasospasm (bilateral with multiple vessel involvement). Parenchymal filling time was calculated as the time delay between initiation of contrast injection till the appearance of parenchymal blush. Venous sinus filling time was calculated as the time delay between the initiation of contrast injection till the appearance of superior sagittal sinus. After diagnosis of vasospasm patients were administered ultrasound guided Stellate Ganglion block using 10 ml of 0.5% Injection Bupivacaine on the same side of vasospasm or the side contralateral to the focal neurological deficit.

Ultrasound Guided Stellate Ganglion Block - Technique Patients were kept supine with the neck in slight hyperextension. Under aseptic conditions, transducer is placed on the surface of the neck at the level of Cervical (C6) vertebrae. The internal jugular vein, carotid artery, thyroid gland, trachea, C6 vertebrae, transverse process of C6, esophagus, longus colli with its covering prevertebral fascia and esophagus are visualized. The transducer was pressed between the trachea and the carotid artery to retract the artery laterally as well as to position the transducer near the longus colli. A 25-gauge Quincke spinal needle was inserted paratracheal towards the middle of the longus colli muscle. The endpoint of the injection was the ultrasound image of the tip of the needle as it penetrates the prevertebral fascia covering the longus colli muscle. The drug is then injected and spread of drug is visualized as distension of prevertebral fascia around the longus colli muscle in real time.

Post Block Assessment-

• Development of ipsilateral Horner Syndrome at 5 minutes interval till 30 minutes after block to confirm successful Stellate Ganglion Block.

At thirty minutes after the block the following parameters are assessed:-

* Neurological condition (GCS score, motor deficits, aphasia, apraxia, hemianopia or neglect). Assessment was done by a blinded neurosurgeon.
* Hemodynamic parameters: heart rate, blood pressure
* Transcranial doppler measurement of flow velocity in MCA, Pulsatility index(PI), Resistivity Index(RI) and LINDEGAARD ratio.
* Digital subtraction angiography was repeated to measure diameter of the vessels affected by vasospasm, change in grading of vasospasm, any increase in vessel diameter, parenchymal filling time and venous sinus filling time. Any increase or decrease in parenchymal and venous sinus filling time was noted.

Block Failure- Block was considered a failure if no signs of Horner's syndrome appeared after 30 minutes of SGB block.

Ineffective Stellate ganglion block- Block was considered ineffective after 30 minutes of Stellate ganglion block

* If there was no neurological improvement
* No improvement in Transcranial doppler findings to normal level or no significant change in affected vessel diameter, grading of vasospasm, parenchymal filling time and venous sinus filling time in second Digital subtraction angiography Rescue Management In case of ineffective block, patients were given intra-arterial nimodipine at rate of 0.1 milligram / minute for a maximum dose of 3 milligram /artery as a rescue measure.

Following this improvement, these patients were monitored in Intensive care unit(ICU).

Management Of Patient In Intensive Care Unit

* Avoidance of hypotension. Maintenance of Systolic Blood Pressure(SBP) at 160-200 mm of Hg using vasopressor {(phenylephrine 2-17microgram/Kg/min) and/or (dopamine-5-10 microgram/kg/min)}
* Avoidance of hypovolemia, maintain Central venous pressure at 8-10 mm of Hg
* Maintenance of Hemoglobin ≥ 9gram/decilitre
* Oral/nasogastric Nimodipine 60mg 4 hourly. Clinical course of patients was followed. Baseline neurological, hemodynamic and TCD parameters were reassessed by the anesthesiologist at 30 minutes . Patients with effective block were reassessed for neurological status and flow velocity measurements by Transcranial Doppler at 6 hours, 12 hours, 24 hours, 36 hours and 48 hours after Stellate ganglion block. Patients with ineffective block who received rescue management were not reassessed for neurological status and flow velocity measurements using Transcranial Doppler at various intervals by the anesthesiologist. However the complications occurring in them, the duration of their stay in the hospital and the final outcome in the form of discharge or death was noted.

Complications Of Stellate ganglion block Procedure and drug-related complications were noted.

Complications During Hospital Stay Complications occurring in the post Stellate Ganglion Block period during the entire hospital stay other than those due to the stellate ganglion block per se were noted. Duration of hospital stay was also noted.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with post aneurysm clipping having symptomatic vasospasm i:e new onset of focal neurological impairment such as hemiparesis, aphasia, apraxia, hemianopia, or neglect or decrease of at least 2 points on the Glasgow Coma Scale (GCS) and duration of symptoms lasting for at least 1 hour.
* Transcranial doppler confirmation of vasospasm by measuring cerebral blood flow velocity in MCA and LINDEGAARD ratio.
* Cerebral angiographic confirmation of the presence of vasospasm by Digital subtraction angiography

Exclusion Criteria:

* New onset of focal neurological deficit or deterioration in the level of consciousness due to other causes like re-bleeding, hydrocephalus, cerebral edema, electrolyte disorder, infection and seizure.
* Patients having an infarct on cerebral tomography.
* Patients with clipping of more than one aneurysm.
* Patients with bilateral neurological deficits.
* History of allergy to local anaesthetic agents.
* Refusal of consent.
* Deranged coagulation profile.
* Patients with pre-existing pupillary changes where assessment of effectiveness of Stellate ganglion block will be difficult.
* History of allergy to contrast media.
* Derangement of renal parameters

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-09; Primary Completion 2015-04 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in Glasgow Coma Scale from baseline that will occur after giving stellate ganglion block in post clipping cerebral vasospasm patients | change in Glasgow Coma Scale from baseline will be assessed a 30 minutes,1 hour, 6,12, 24, 36, 48 hours
Change in motor power on motor system examination from baseline that will occur after giving stellate ganglion block in post clipping cerebral vasospasm patients | change in motor power on motor system examination from baseline will be assessed a 30 minutes,1 hour, 6,12, 24, 36, 48 hours
Presence or absence of aphasia before and after stellate ganglion block | it will be assessed at baseline and 30 minutes,1 hour, 6,12, 24, 36, 48 hours after stellate ganglion block

SECONDARY OUTCOMES:
Change in Peak systolic velocity on Transcranial doppler from baseline that will occur after giving stellate ganglion block in post clipping cerebral vasospasm patients | Parameters will be assessed at Baseline and 30 minutes,1 hour, 6,12, 24, 36, 48 hours after the block
Change in Mean Flow Velocity on Transcranial Doppler from baseline that will occur after giving stellate ganglion block in post clipping cerebral vasospasm patients | Parameters will be assessed at Baseline and 30 minutes,1 hour, 6,12, 24, 36, 48 hours after the block
Change in LINDEGAARD ratio on Transcranial Doppler from baseline that will occur after giving stellate ganglion block in post clipping cerebral vasospasm patients | Parameters will be assessed at Baseline and 30 minutes,1 hour, 6,12, 24, 36, 48 hours after the block
Change in Pulsatility Index on Transcranial Doppler from baseline that will occur after giving stellate ganglion block in post clipping cerebral vasospasm patients | Parameters will be assessed at Baseline and 30 minutes,1 hour, 6,12, 24, 36, 48 hours after the block
Change in vessel calibre on Digital Subtraction Angiography from baseline that will occur after giving stellate ganglion block in post clipping cerebral vasospasm patients | Parameters will be assessed at Baseline and 30 minutes
Change in parenchymal filling time on Digital Subtraction Angiography from baseline that will occur after giving stellate ganglion block in post clipping cerebral vasospasm patients | Parameters will be assessed at Baseline and 30 minutes
Change in Venous sinus filling time on Digital Subtraction Angiography from baseline that will occur after giving stellate ganglion block in post clipping cerebral vasospasm patients | Parameters will be assessed at Baseline and 30 minutes

IPD SHARING:
Plan to Share IPD: Undecided